CLINICAL TRIAL: NCT05728164
Title: The Power of Cinematic Simulation as Action to Regulate Emotions, Leverage Resilience, and Foster Empathy Among Undergraduate Nursing Students: A Randomized Control Trial
Brief Title: Effect of Cinematic Simulation on Emotions, Resilience, and Empathy Among Undergraduate Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1022013
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Power of Cinematic Simulation on Emotions, Resilience, and Empathy Among Undergraduate Nursing Students

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): The group (35 students) will be divided into 7 small groups of (5 students in each group). In addition to routine training provided for the control group, the students of the intervention group will be provided with micro learning content following the educational topics of the course in the form of short videos of cinematic films reinforcing values of resilience, empathy, and positive emotions in dealing with others.
  • Pre-simulation activities will also be developed that required watching a tutorial video on how to create a plan of care for such cases. Students also will be provided with background on cinematic simulation and a summary of the characters. Learners will be assigned to one of the films characters and introduced to the assessment tool they would utilize. A pre-briefing discussion on patient confidentiality, nursing role expectations, and developing a plan of care also preceded the activity.
  Interventions: Behavioral: Cinematic Simulation
- Cintrol group (No Intervention): They will receive usual training based on the educational objectives of routine methods of lectures, discussion.

INTERVENTIONS:
Behavioral: Cinematic Simulation — Comprehensive videos from specific films will be selected as films fitting the needs of participants and the established objectives. The films comprehensively develops several characters enriching the values of positive emotions, resilience and empathy. The intervention film videos will be delivered on 5 sessions for each group (2 sessions per week).
  Arms: STUDY GROUP

SUMMARY:
The aim of this study is to:

Determine the effect of cinematic simulation as action to regulate emotions, leverage resilience, and foster empathy among undergraduate nursing students.

Research Hypothesis Nursing students who participated in cinematic simulation will exhibit better regulation of emotions, resilience, and empathy than those in the control group

DETAILED DESCRIPTION:
The current study's population was the second-term "4th level" registered undergraduate nursing candidates in the year 2022/2023.

A sample of 70 randomly selected students from the psychiatric nursing rotation will be included in this study. The study subjects will be divided equally into two groups (study and a control group) matched as much as possible. The exclusion criteria include students who were not willing to participate in the study, those who complained of any mental disorders or had a previous history of any mental problems.

Assigned students will be randomly divided into two groups of intervention; study (n = 35) and control (n = 35). The control group will receive usual training based on the educational objectives of routine methods of lectures, discussion, …etc.

The study group (35 students) will be divided into 7 small groups of (5 students in each group). In addition to routine training provided for the control group, the students of the intervention group will be provided with micro learning content following the educational topics of the course in the form of short videos of cinematic films reinforcing values of resilience, empathy, and positive emotions in dealing with others.

Objectives for the cinematic simulation included the following: 1) apply the principles of positive emotions, empathetic understanding and resilience to students from diverse backgrounds; 2) analyze the care management process as it relates to assessment, goals, interventions, teaching, and outcomes in mental health nursing; and 3) Reinforcing the psychological role of the professional nurses in caring for patients with different diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian Nursing students

Exclusion Criteria:

complained of any mental disorders or had a previous history of any mental problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire: | 2 weeks
  The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report scale designed to assess habitual use of two commonly used strategies to alter emotion: cognitive reappraisal and expressive suppression. Participants respond to each item using a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Cognitive reappraisal involves thinking differently about a situation in order to change its meaning in order to alter one's emotional experience.

SECONDARY OUTCOMES:
The Connor-Davidson Resilience Scale | 2 weeks
  The Connor-Davidson Resilience Scale (CD-RISC) is a test that measures resilience, or readiness to bounce back after a stressful event, tragedy, or trauma. It consists of 25 items, each rated on a 5-point scale (0-4), as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all the time (4). Reliability, validity, and factor analysis structure of scales were assessed and reference values for study samples were calculated. The ratings result in a number between 0-100, and higher scores indicate higher resilience. Scores are categorized as follows: < 50% for low resilience levels and ≥50% for high resilience levels.

OTHER OUTCOMES:
Toronto Empathy Questionnaire (TEQ) | 2weeks
  The Toronto Empathy Questionnaire was constructed by (Spreng), 2009. TEQ is a 16-item (eight items are scored negatively and eight items are scored positively) on five-point Likert type scale. The scale assesses the frequency that the statements are considered true and ranges from 0 = never, 1 = rarely, 2 = sometimes, 3 = often to 4 = always)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No